CLINICAL TRIAL: NCT06093516
Title: The ARUTIS Study (Anglia Ruskin University Trial of the Intuitive System) A Single-centre, Double-masked Randomised Controlled Crossover Trial of Precision Tinted Lenses for Visual Stress
Brief Title: The ARUTIS Study (Anglia Ruskin University Trial of the Intuitive System)
Acronym: ARUTIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anglia Ruskin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ETH2223-7100
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-09

CONDITIONS: Visual Stress
Keywords: Visual stress; Intuitive system; Intuitive colorimeter; Colorimetry; Precision Tinted Lenses; Wilkins Rate of Reading test

STUDY DESIGN:
Intervention Model Description: The ARUTIS study is a double-masked randomised controlled trial (RCT) having a double-masked crossover (AB/BA) design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Optimal Precision Tinted Lenses (PTL) (Experimental): 1. The participant is asked to describe any perceptual distortion and discomfort of the text in the colorimeter.
  2. At each of the 12 hues in turn the saturation of colour is increased from white to modest saturation (30) and after 5s returned to white. The participant is asked to compare the coloured text with the white and report any differences in the distortion/discomfort.
  3. At the best of the 12 hues, the participant adjusts the saturation to optimise the clarity and comfort of the text (comfort is more important than clarity).
  4. At this saturation, the hue is adjusted by small amounts and re-optimised. The saturation is then minimised.
  5. At the re-optimised hue/saturation, the brightness is reduced to assess its effects on comfort. If the lower brightness is preferred the saturation is increased slightly to see if the high brightness is better tolerated.
  Interventions: Device: Tinted Lenses
- Sub-Optimal Precision Tinted Lenses (PTL) (Experimental): The sub-optimal colour will be chosen as a colour of similar saturation to the optimal colour but differing in u'v' colour space by 0.07. Two colours of equal radial distance from the optimal colour will be considered. The colour that shares the name of the optimal colour or appears most similar will be chosen.
  After colorimetry, participants will choose a spectacle frame. Two pairs of PTLs will be made up by the manufacturing opticians, one to the optimal colour and the other to a slightly sub-optimal colour.
  Interventions: Device: Tinted Lenses

INTERVENTIONS:
Device: Tinted Lenses — Tinted coloured lenses with UV protection within spectacle frames with the intension to help reduce the symptoms of Visual stress.

SUMMARY:
The goal of this double-masked randomised controlled trial (RCT) is to assess the symptoms of visual stress (VS), reading speed and changes in behaviour / academic performance, when wearing optimal Precision Tinted Lenses compared to sub-optimal Precision Tinted Lenses (PTLs). In participants ages 9-18 years.

Participants, parents and researchers will be masked until the end of the trial.

Participants will be randomised into two groups A and B. 50% of participants will receive the optimal PTL where the other 50% will receive the sub-optimal PTL.

Participants will be asked to wear the PTLs for one month. Followed by one month of no wear. After which, participants will receive the second pair of PTLs to wear for one month.

Participants will need to fill out a symptom dairy everyday from the day of recruitment until the end of the trial. A symptom questionnaire will need to be filled out as baseline at recruitment and the end of each month of wear. An academic behaviour survey will also need to be filled out at baseline by parents and teachers at recruitment and the end of each month of wear.

At the end of the three months unmasking will occur and participants will be given the PTL that demonstrate the greatest reduction in VS.

DETAILED DESCRIPTION:
The ARUTIS study is a double-masked randomised controlled trial (RCT) having a double-masked crossover (AB/BA) design. The study aims to assess the symptoms of visual stress (VS), reading speed and changes in behaviour / academic performance, when wearing optimal Precision Tinted Lenses compared to sub-optimal Precision Tinted Lenses (PTL). The PTLs will be prescribed by the Intuitive System.

A total of 120 participants aged 9-18 years with symptoms of VS will be recruited from the Anglia Ruskin University eye clinic. Participants will be randomised into either Group 1 (receiving the two interventions A (optimal tint) and B (sub-optimal) in the order AB) or Group 2 (receiving the two interventions in the order BA).

The initial pair of PTLs will be given to participants for a one-month wearing period. Subsequently, a one-month washout period is observed, after which participants receive the second pair of PTLs for one-month. Participants are required to fill out a symptom diary daily. A symptom questionnaire will need to be filled out as baseline at recruitment and the end of each month of wear. An academic behaviour survey will also need to be filled out at baseline by parents and teachers at recruitment and the end of each month of wear. Following the three months, a head-to-head comparison and unmasking will occur.

Participants will be given the Precision Tinted Lenses that demonstrate the greatest reduction in VS. The study will combine quantitative and qualitative data collection. The primary outcome measure is comparing symptom scores with questionnaires and symptom diaries reported under two different treatment conditions. The secondary outcome measures will be evaluated. in two ways: change in reading speed and results from academic behaviour surveys.

ELIGIBILITY:
Inclusion Criteria:

1. Age 9-18y.
2. Meet diagnostic indicators for visual stress (see below)
3. Consent (parent and participant to attend for optometric testing and participate in research.
4. Do not anticipate moving from the area in the next 3 months

Diagnostic indicators for visual stress

At least three of the following six typical symptoms:

1. Words Move
2. Words Merge
3. Patterns or shadows in text (e.g., "rivers")
4. Text seems to stand out in 3-D above the page
5. Words or letters fade or darken
6. Discomfort with certain artificial lights and flicker

And "At least two of the following three signs from investigations:

1. Voluntary unprompted use of an overlay for 3 months or more
2. Overlay improves performance at the WWRT BY ≥15%
3. PGT result >3 with mid spatial frequency grating.

Exclusion Criteria:

1. History of wearing precision tinted lenses.
2. Ocular pathology, systemic pathology that is likely to worsen in the timescale of the study or cause transient blur (e.g., diabetes) or photosensitive epilepsy

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-10-30 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Comparing symptom scores with symptom diaries reported under the two different treatment conditions | 3 months
  Participants will be requiured to fill out a daily diary from day of recruitment to the end of the trial.
Comparing symptom scores with questionnaires reported under the two different treatment conditions. | 3 months
  Participants will be required to fill out symptom questionnaires at baseline and at the end of each month wear.

SECONDARY OUTCOMES:
Identify the change in reading speed for participants (if any) when wearing PTLs, by analysing the results of the Wilkins Rate of Reading test (WRRT). | 3 months
  Participants will be required to perform a WRRT at baseline and at the collection of each PTLs.
  A WRRT will also be performed at the unmasking stage to compare both PTLs.
Identify the academic/behavioural change (if any) in participants when wearing PTLs, by analysing a survey completed by parents/guardians and teachers. | 3 months
  Parents/ teachers will be required to fill out the the academic/behavioural survey at baseline and at the end of each month wear.

CONTACTS AND LOCATIONS:
Locations (1):
- Anglis Ruskin University, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The study will conform to the tenets of the Declaration of Helsinki and will be registered in a clinical trials registry. When the analysis is complete, anonymised data will be stored in a publicly accessible data repository. Full informed consent will be obtained from participants and parents/guardians. Ethical approval was granted from the Anglia Ruskin University Faculty Research Ethics Panel (FREP).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available after the trial has been completed. Which will be in approximately 12 months.
  Data will be available for as long as necessary.